CLINICAL TRIAL: NCT02581982
Title: Single-Arm Phase II Combination Study of Low-Dose Paclitaxel With Pembrolizumab in Platinum-Refractory Urothelial Carcinoma
Brief Title: Paclitaxel and Pembrolizumab in Treating Patients With Refractory Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00035397; NCI-2015-01713 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 88215 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Transitional Cell Carcinoma
Keywords: Urothelial cancer; Bladder cancer; Immunotherapy; Paclitaxel
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, paclitaxel) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and paclitaxel IV over 60 minutes on day 1 and 8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well paclitaxel and pembrolizumab works in treating patients with urothelial cancer that has not responded to previous treatment and has spread to other places in the body. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Giving paclitaxel together with pembrolizumab may be an effective treatment for urothelial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall response rate (ORR) of pembrolizumab combined with paclitaxel.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of pembrolizumab combined with paclitaxel.

II. To calculate the progression-free survival (PFS) rate at 6 months.

TERTIARY OBJECTIVES:

I. To determine the immune effects of pembrolizumab combined with paclitaxel. II. To associate immune effects with tumor response. III. To explore changes in immune-regulatory micro ribonucleic acids (RNAs) as biomarkers of response.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and paclitaxel IV over 60 minutes on day 1 and 8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with platinum-refractory metastatic urothelial cancer that is measureable based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1.36 Platinum-refractory disease is defined as progressive disease on cisplatin or carboplatin therapy or within 12 months of prior platinum treatment (last dose.)
* At least 1 prior chemotherapy regimen containing cisplatin or carboplatin
* Patient must be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 months (168 days) prior to initiation of treatment on Day 1. Archived specimen can be used for subjects, if available
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Adequate organ function as defined below:
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 80,000 / mcL
* Hemoglobin >= 9 g/dL without transfusion dependency
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance rate [CrCl]) >= 35 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Currently receiving or has had treatment with an investigational agent or used an investigational device within 4 weeks of study day 1
* Anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death-ligand 1 (PD-L1), or anti-programmed cell death-ligand 2 (PD-L2) agent. Prior therapy with paclitaxel or docetaxel
* Hypersensitivity to pembrolizumab, any of its excipients, paclitaxel, or any of its excipients
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Known history of active TB (Bacillus tuberculosis)
* Known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known history of, or any evidence of active, non-infectious pneumonitis
* Active infection requiring systemic therapy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnancy or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goodman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Paclitaxel)
Started | 27
Completed | 11
Not Completed | 16
Not completed — Lack of Efficacy | 12
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Paclitaxel)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 21
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The overall response rate will be performed in all patients that are evaluable for efficacy and will have one interim analysis. Overall response is complete response (CR) = Disappearance of all target lesions (PR) = at least a 30% decrease in sum of diameters, taking as reference the baseline sum diameters; stable disease (SD) = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum diameters while on study; and progressive disease (PD) = at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study based on all target lesions recorded since the treatment started.
Time Frame: Up to 6 months
Population: Out of the 27 participants, only 25 were evaluable for response to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Paclitaxel)
Number analyzed (Participants) | 25
Participants
  Complete Response | 3
  Partial Response | 6
  Stable Disease | 9
  Progressive Disease | 7

2. Secondary Outcome: Number of Adverse Events Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: All adverse events will be tabulated and presented by preferred term and/or system organ class and grade. All deaths and serious adverse events will be tabulated.
Time Frame: Up to 1 year
Measure: Number; unit: Adverse Events
Arm/Group | Treatment (Pembrolizumab, Paclitaxel)
Number analyzed (Participants) | 27
Adverse Events
  Serious adverse events | 34
  Adverse events | 61

3. Secondary Outcome: Progression Free Survival (Kaplan Meier Method)
Description: The Kaplan Meier methods will be used to estimate progression free survival. The 6-month PFS will be compared to historical rates using a chi-square test. Progressive disease is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study based on all target lesions recorded since the treatment started. The sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression)
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, Paclitaxel)
Number analyzed (Participants) | 27
percentage of participants | 44 [26 to 62]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Pembrolizumab, Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 4/27
Serious Adverse Events (participants affected / at risk) | 27/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Paclitaxel) (N=27)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Death (General disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypethyroidism (Endocrine disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 1 (1) — Duodenitis
Renal and urinary disorders - other (Renal and urinary disorders) | 1 (1) — Pyelonephritis
Surgical and medical procedures - other (Surgical and medical procedures) | 1 (1) — Intramedullary rod placement of tibia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Paclitaxel) (N=27)
Abdominal pain (Gastrointestinal disorders) | 7 (8)
Alanine aminotransferase increased (Investigations) | 4 (9)
Alkaline phosphatase increased (Investigations) | 7 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (24)
Anemia (Blood and lymphatic system disorders) | 20 (96)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 7 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Chills (General disorders) | 5 (6)
Chronic kidney disease (Renal and urinary disorders) | 13 (61)
Constipation (Gastrointestinal disorders) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (15)
Creatinine increased (Investigations) | 10 (36)
Diarrhea (Gastrointestinal disorders) | 4 (13)
Dizziness (Nervous system disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Edema limbs (General disorders) | 4 (9)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 21 (66)
Fever (General disorders) | 5 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (7)
Hematuria (Renal and urinary disorders) | 7 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (70)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4)
Hypertension (Vascular disorders) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (48)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (13)
Hypokalemia (Metabolism and nutrition disorders) | 6 (16)
Hypomagenesemia (Metabolism and nutrition disorders) | 7 (8)
Hyponatremia (Metabolism and nutrition disorders) | 12 (23)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (8)
Infusion related reaction (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (22)
Lymphedema (Vascular disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 15 (42)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 12 (23)
Neutrophil count decreased (Investigations) | 4 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 6 (16)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (10)
Platelet count decreased (Investigations) | 9 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (13)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (7)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 16 (48)
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 2 (4) — Rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT02581982/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT02581982/ICF_001.pdf